CLINICAL TRIAL: NCT04527887
Title: Intracanalicular Dexamethasone Insert for the Treatment of Inflammation and Discomfort in Dry Eye Disease
Brief Title: Intracanalicular Dexamethasone Insert for the Treatment of Inflammation and Discomfort in Dry Eye Disease (DEcIDED)
Acronym: DEcIDED
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Per sponsor decision due to lengthy enrollment period
Sponsor: Tufts Medical Center (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00000084
Record Dates: First submitted 2020-02-19; First posted 2020-08-27 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dextenza (IDI) (Sustained Release Dexamethasone, (0.4 mg) (Active Comparator): intracanalicular dexamethasone insert
  Interventions: Drug: Dextenza (IDI) (Sustained Release Dexamethasone), (0.4 mg)
- ProLong™ collagen plugs (Placebo Comparator): collagen plug
  Interventions: Other: ProLong™ collagen plugs

INTERVENTIONS:
Drug: Dextenza (IDI) (Sustained Release Dexamethasone), (0.4 mg) — Intracanalicular dexamethasone insert contains 0.4 mg dexamethasone and is designed to provide a sustained and tapered release of therapeutic levels of dexamethasone to the ocular surface for up to 30 days for the reduction of postsurgical inflammation and pain associated with ocular surgery.
  Arms: Dextenza (IDI) (Sustained Release Dexamethasone, (0.4 mg)
Other: ProLong™ collagen plugs — The long term synthetic punctal plug is composed of an absorbable copolymer material and measures 0.4mm in diameter and 2.0mm in length.
  Arms: ProLong™ collagen plugs

SUMMARY:
This prospective, single-center, randomized, double-masked, parallel comparison, sponsored study seeks to investigate the efficacy of Intracanalicular dexamethasone Insert (IDI) on ameliorating the signs and symptoms of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Dry Eye Disease
* Objective Signs (Schirmer's II test <10 mm at 5 min; Tear Break-Up time (TBUT) of <10 seconds in 1 eye; corneal fluorescein staining of .=4 in at least 1 eye; conjunctival lissamine green staining of the nasal and temporal conjunctive >=4 in at least 1 eye)
* Ocular inflammation presence confirmed by In-Vivo Confocal Microscopy

Exclusion Criteria:

* History of Diabetes
* History of ocular surgery, corneal infection, or corneal injury within the last 3 months
* Active ocular allergies
* Active ocular infection
* Allergic to benzalkonium chloride

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in ocular inflammation | Change from Baseline one month after intracanalicular insert implantation or punctal plug
  As measured by change to dendritic cell density and ocular redness

SECONDARY OUTCOMES:
Clinical Parameter: Ocular Surface Disease Index (OSDI) | Change from Baseline one month after intracanalicular insert implantation or punctal plug
  12-item scale; score ranges from 0 to 100 and is calculated by the sum of the scores for all 12 questions answered multiplied by 100, which is divided by the total number of questions answered times four
Clinical Parameter: Ocular Pain Assessment Survey (OPAS) | Change from Baseline one month after intracanalicular insert implantation or punctal plug
  32-questions, 8-domain questionnaire using numerical rating scales to assess eye pain intensity (worse eye) in the past 24 hours and 2 weeks (worst, least and average pain intensity), frequency of eye and non-eye pain (past 24 hours and 2 weeks), non-eye pain intensity (past 24 hours and 2 weeks), impact on QoL, pre-occupation with eye and non-eye pain, aggravating factors and associated factors.)
Clinical Parameter: Symptom Assessment in Dry Eye scores (SANDE) | Change from Baseline one month after intracanalicular insert implantation or punctal plug
  Score is calculated by multiplying the frequency of symptoms score with the severity of symptoms score and obtaining the square root.
Clinical Parameter: Tear Break Up Time (TBUT) | Change from Baseline one month after intracanalicular insert implantation or punctal plug
  The standard TBUT measurement will be performed by dropping a fluorescein drop to the inferior tarsal conjunctiva and waiting 30 seconds. After several blinks, the tear film will be examined. The time lapse between the last blink and the appearance of the first randomly distributed dark discontinuity in the fluorescein stained tear film will be measured three times and the mean value of the measurements will be calculated.
Clinical Parameter: Conjunctival staining | Change from Baseline one month after intracanalicular insert implantation or punctal plug
  Grading of conjunctival lissamine green staining will be performed after 1 minutes of application of a lissamine green drop. Staining will be graded using the National Eye Institute (NEI) grading scheme, with a total range of 0-18.
Clinical Parameter: Corneal staining with fluorescein | Change from Baseline one month after intracanalicular insert implantation or punctal plug
  Corneal fluorescein staining will be performed after 2 minutes of application of a fluorescein drop. Staining will be graded using the National Eye Institute (NEI) grading scheme, with a total range of 0-15.
Clinical Parameter: Schirmer II test | Change from Baseline one month after intracanalicular insert implantation or punctal plug
  Aqueous tear production will be measured by the length in millimeters that the strip wets during 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Hamrah, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No